CLINICAL TRIAL: NCT01251549
Title: Safety and Performance Evaluation of ReWalk Reciprocating Gait Orthosis (RGO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ReWalk Robotics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RW003 ver. 4
Record Dates: First submitted 2010-11-28; First posted 2010-12-02 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Paraplegia; Spinal Cord Injuries (SCI)
Keywords: ReWalk; Paraplegia; Spinal Cord Injuries (SCI)
MeSH Terms: conditions — Paraplegia; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental: A (Experimental): A group of paraplegics.
  Interventions: Device: ReWalk - a motorized exoskeleton suit

INTERVENTIONS:
Device: ReWalk - a motorized exoskeleton suit — The subject will wear the ReWalk suit and have training sessions for walking with the device
  Other Names: Exoskeleton suit

SUMMARY:
ReWalk suit developed by Argo Medical Technologies is designed to enable people with lower limb disabilities to carry out routine ambulatory functions (stand, walk etc.); it can be used by people with disabilities such as spinal cord injury, brain injury, stroke, multiple sclerosis, cerebral palsy and other pathologies that produce severe walking impairments.

ELIGIBILITY:
Inclusion Criteria:

* Complete cervical (C7-8) or thoracic (T1-T12) spinal cord injury according to American Spinal Injury Association (ASIA) guidelines
* Male and non-pregnant non-lactating female Age 18-55
* At least 6 months after injury
* Regular use of RGO (Reciprocating Gait Orthosis) or KAFO's (Knee Ankle Foot Orthoses) or able to stand using a standing device (e.g., 'Easy stand')
* Patients must be capable of providing informed consent
* Height of 160 to 190 cm
* Weight of <100 kg

Exclusion Criteria:

* History of severe neurological injuries other than SCI (Spinal Cord Injuries)(MS (Multiple Sclerosis), CP (Cerebral Palsy), ALS (Amyotrophic Lateral Sclerosis) , TBI (Traumatic Brain Injury) etc)
* Severe concurrent medical diseases: infections, circulatory, heart or lung, pressure sores
* Severe spasticity (Ashworth 4) or uncontrolled clonus
* Unstable spine or unhealed limbs or pelvic fractures
* Heterotopic ossification
* Significant contractures
* Psychiatric or cognitive situations that may interfere with the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety of use | 3 months
  Number of participants with related adverse events as a Measure of Safety and Tolerability

SECONDARY OUTCOMES:
Efficacy | 3 months
  Continuously walking for 6 minutes after 18 sessions training with the ReWalk - exoskeleton suit performed at weekly intervals

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Esquenazi, MD, Principal Investigator — Albert Einstein Medical Center, Moss Rehabilitation Center
Locations (2):
- Albert Einstein Medical Center, Moss Rehabilitation Center, Elkins Park, Pennsylvania, United States
- Ospedale Valduce di Como, Centro Villa Beretta Italy, Como, Italy